CLINICAL TRIAL: NCT03552354
Title: Argatroban Combined With Antiplatelet Versus Antiplatelet for Acute Mild or Moderate Ischemic Stroke With Large-artery Atherosclerosis: a Prospective, Single Center Study
Brief Title: Argatroban Combined With Antiplatelet Versus Antiplatelet for Acute Ischemic Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director of the Department, General Hospital of Shenyang Military Region
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: k(2017)38
Record Dates: First submitted 2018-04-27; First posted 2018-06-11 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — argatroban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Argatroban combined with antiplatelet (Experimental)
  Interventions: Drug: Argatroban plus dual antiplatelet

INTERVENTIONS:
Drug: Argatroban plus dual antiplatelet — A continuous argatroban infusion of 1.0 ug/kg per minute for 2-5 days adjusted to a target activated partial thromboplastin time of 1.75 X baseline (about 10%). For the first day, clopidogrel with loading dose 300mg, and aspirin 100mg were given, and followed by clopidogrel 75 mg and aspirin 100mg each day

SUMMARY:
Intravenous thrombolysis is considered as the first choice for ischemic stroke. In the recent years, endovascular therapy is demonstrated to be effective to treat ischemic with big vessel occlusion. However, only a minority of patients can get intravenous thrombolysis or endovascular therapy due to the restricted time window and strict indications. Dual antiplatelet has been demonstrated to be effective in the patients with high risk of TIA or minor ischemic stroke (NIHSS<4). But there is still stroke progression although dual antiplatelet. The ischemic stroke patients with NIHSS > 3 has been recommended to give aspirin in most guidelines. Of those patients, mild to moderate stroke patients (3<NIHSS<10) will result in the poor outcomes if the progression occurs. In addition, large artery atherosclerosis (LAA) stroke is prone to progress. So, we argue that the mild to moderate stroke with LAA should be give more intensive antiplatelet. In the present study, argatroban combined with antiplatelet therapy (3-5 days) is used to treat the proposed patients to investigate the safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old;
2. Clear diagnosis of ischemic stroke patients with head CT or MRI examination;
3. The time of onset is less than 72 hours;
4. NIHSS score is less than 12 points;
5. the large artery atherosclerosis etiology
6. Signed informed consent.

Exclusion Criteria:

1. Hemorrhagic stroke or mixed stroke;
2. Patients with planned thrombolytic therapy;
3. Serious diseases such as severe infection or liver, kidney, hematopoietic system, endocrine system, etc.;
4. The history of stroke and had serious sequelae (mRS> 1);
5. Allergic to aspirin/clopidogrel and argatroban;
6. ischemic stroke caused by other causes, such as small vessel lesions, cardiogenic embolism, arterial dissection, vasculitis and other cerebral infarction;
7. Previous history of cerebral hemorrhage;
8. It is expected to use other anti-platelet agents or non-steroidal anti-inflammatory agents that affect platelet function;
9. within 3 months of gastrointestinal bleeding or major surgery;
10. any unqualified patients judged by researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Proportion of 1 or more increase in NIHSS | 7 days
  early neurological deterioration is defined as 1 or more increase in NIHSS

OTHER OUTCOMES:
Proportion of mRS 0-1 | 90±7 days
  the excellent outcome is defined as modifed Rankin Score (mRS) 0-1 at 90 day
Proportion of mRS 0-2 | 90±7 days
  the good outcome is defined as modifed Rankin Score (mRS) 0-2 at 90 day
proportion of intracranial haemorrhages | 90±7 days
  intracranial hemorrhage was defined as acute extravasation of blood into the brain parenchyma or subarachnoid space with associated neurologic symptoms
proportion of organs hemorrhage | 90±7 days
  including gastrointestinal bleeding and mucocutaneous hemorrhage
death | 90±7 days
  death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Shenyang Military Region, Shenyang, Liaoning, China